CLINICAL TRIAL: NCT03134560
Title: Comparison Between Using Vein Display Instrument and Without Using Vein Display Instrument for Successful Intravenous Cannulation in Pediatric Patients
Brief Title: Intravenous Cannulation Using Vein Display Instrument and Without Using Vein Display Instrument in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aries Perdana, Consultant, Anesthesiologist, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes003
Record Dates: First submitted 2017-04-24; First posted 2017-05-01 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Difficult Vein Access
Keywords: vein display instrument; pediatric; vein access; vein cannulation

ARMS (2):
- With vein display instrument (Active Comparator): Vein cannulation was done after the vein display instrument displays the veins using infrared
  Interventions: Device: Vein Display Instrument
- Without vein display instrument (No Intervention): vein cannulation was done without any vein display instrument

INTERVENTIONS:
Device: Vein Display Instrument
  Arms: With vein display instrument

SUMMARY:
This study aims to compare intravenous cannulation success rate between using vein display instrument and without using vein display instrument in pediatric patients.

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Parents' subjects were given informed consent before enrolling the study. After doing asepsis and antisepsis procedure and putting on the tourniquet the first group would get intravenous cannulation without vein displaying instrument. While for the second group, after doing asepsis procedure and tourniquet was put on, a vein display instrument was used to choose the vein. Intravenous cannulation was done after antiseptic procedure. After blood dripped out of the cannula, cannula was connected to the infusion set. Evaluation was done to assess vein route establishment, canulation attempt number and swelling. Data recorded were analyzed using Statistical Package for the Social Sciences (SPSS) using Chi-square test or Fisher Exact test. Significant value is p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 0-5 years old
* Subjects with difficult vein access (e.g. edema, obesity, chemotherapy history),
* Subjects whose parents had signed the informed consent
* Subjects with available vein access locations at the back of either hands.

Exclusion Criteria:

* Subjects who had infection signs at the designated vein access location
* Subjects in need of emergency procedures.

Drop out Criteria:

* Subjects resigned from the study
* Subjects rejected any next attempt of intravenous cannulation
* Subjects who received anesthetic drugs before intravenous cannulation.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2016-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Successful first vein cannulation attempt | Day 1
  Whether the first vein cannulation attempt successful or not will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Aries Perdana, Consultant, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Myers LA, Arteaga GM, Kolb LJ, Lohse CM, Russi CS. Prehospital peripheral intravenous vascular access success rates in children. Prehosp Emerg Care. 2013 Oct-Dec;17(4):425-8. doi: 10.3109/10903127.2013.818180. Epub 2013 Aug 16. PMID 23952007
- [Background] Scales K. Vascular access: a guide to peripheral venous cannulation. Nurs Stand. 2005 Aug 17-23;19(49):48-52. doi: 10.7748/ns2005.08.19.49.48.c3935. PMID 16134420
- [Background] Doniger SJ, Ishimine P, Fox JC, Kanegaye JT. Randomized controlled trial of ultrasound-guided peripheral intravenous catheter placement versus traditional techniques in difficult-access pediatric patients. Pediatr Emerg Care. 2009 Mar;25(3):154-9. doi: 10.1097/PEC.0b013e31819a8946. PMID 19262420
- [Background] Simhi E, Kachko L, Bruckheimer E, Katz J. A vein entry indicator device for facilitating peripheral intravenous cannulation in children: a prospective, randomized, controlled trial. Anesth Analg. 2008 Nov;107(5):1531-5. doi: 10.1213/ane.0b013e318185cdab. PMID 18931210
- [Background] Chapman LL, Sullivan B, Pacheco AL, Draleau CP, Becker BM. VeinViewer-assisted Intravenous catheter placement in a pediatric emergency department. Acad Emerg Med. 2011 Sep;18(9):966-71. doi: 10.1111/j.1553-2712.2011.01155.x. Epub 2011 Aug 19. PMID 21854488
- [Background] Schindler E, Schears GJ, Hall SR, Yamamoto T. Ultrasound for vascular access in pediatric patients. Paediatr Anaesth. 2012 Oct;22(10):1002-7. doi: 10.1111/pan.12005. PMID 22967159
- [Background] Donaldson JS. Pediatric vascular access. Pediatr Radiol. 2006 May;36(5):386-97. doi: 10.1007/s00247-006-0118-1. Epub 2006 Mar 15. PMID 16538464
- [Background] de Negri DC, Avelar AF, Andreoni S, Pedreira Mda L. Predisposing factors for peripheral intravenous puncture failure in children. Rev Lat Am Enfermagem. 2012 Nov-Dec;20(6):1072-80. doi: 10.1590/s0104-11692012000600009. English, Portuguese, Spanish. PMID 23258720
- [Background] Lamperti M, Pittiruti M. II. Difficult peripheral veins: turn on the lights. Br J Anaesth. 2013 Jun;110(6):888-91. doi: 10.1093/bja/aet078. No abstract available. PMID 23687310
- [Background] Kim MJ, Park JM, Rhee N, Je SM, Hong SH, Lee YM, Chung SP, Kim SH. Efficacy of VeinViewer in pediatric peripheral intravenous access: a randomized controlled trial. Eur J Pediatr. 2012 Jul;171(7):1121-5. doi: 10.1007/s00431-012-1713-9. Epub 2012 Mar 14. PMID 22415409
- [Background] Chiao FB, Resta-Flarer F, Lesser J, Ng J, Ganz A, Pino-Luey D, Bennett H, Perkins C Jr, Witek B. Vein visualization: patient characteristic factors and efficacy of a new infrared vein finder technology. Br J Anaesth. 2013 Jun;110(6):966-71. doi: 10.1093/bja/aet003. Epub 2013 Feb 5. PMID 23384732
- [Background] Kaddoum RN, Anghelescu DL, Parish ME, Wright BB, Trujillo L, Wu J, Wu Y, Burgoyne LL. A randomized controlled trial comparing the AccuVein AV300 device to standard insertion technique for intravenous cannulation of anesthetized children. Paediatr Anaesth. 2012 Sep;22(9):884-9. doi: 10.1111/j.1460-9592.2012.03896.x. Epub 2012 Jun 14. PMID 22694242
- [Background] John JM. Transillumination for vascular access: old concept, new technology. Paediatr Anaesth. 2007 Feb;17(2):197-8. doi: 10.1111/j.1460-9592.2006.02061.x. No abstract available. PMID 17238901
- Available data/document: Textbook — https://books.google.co.id/books/about/Pediatric_Anesthesia.html?id=RYe4GBD6LrQC&redir_esc=y — Hannallah RS , Verghese ST. Peripheral vascular access. In: Bissonnette B, Anderson BJ, Bosenberg A, Engelhardt T, Mason LJ, Tobias JD, editors. Pediatric Anesthesia. Connecticut: People's Medical Publishing House USA, 2011.p. 1097-102.